CLINICAL TRIAL: NCT06062914
Title: Health Economic Research on Oral Nutritional Supplements for Hospitalized Patients With Nutritional Risk
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CAJJ-003
Record Dates: First submitted 2023-09-18; First posted 2023-10-02 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Malnutrition; Nutritional Risk
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- oral nutritional supplement group: Only oral nutritional supplement was used as enteral nutrition, including but not limited to Ensure®, Nutrison® and etc.
  Interventions: Drug: oral nutritional supplements
- no-oral nutritional supplement group: no enteral nutrition was received

INTERVENTIONS:
Drug: oral nutritional supplements — Only ONS was used as enteral nutrition
  Groups: oral nutritional supplement group

SUMMARY:
The goal of this observational study is to evaluate the treatment effect and health economic impact of oral nutritional supplements(ONS) in hospitalized patients with nutritional risk. The main questions it aims to answer are:

* To evaluate the effect of ONS on clinical outcomes in hospitalized patients with high nutritional risk
* To evaluate the health economic impact of ONS in hospitalized patients with high nutritional risk Data was collected from patients admitted to peking union medical college hospital between January 1, 2018 and December 31, 2020.

The inclusion criteria were as follows: (1) age≥18 years old; (2)length of hospital stay≥3days; (3) Only ONS was used as enteral nutrition or no enteral nutrition was received.

Exclusion criteria were: (1) age<18; (2) length of hospital stay<3 days; (3) the patients who received enteral nutrition other than ONS (such as tube feeding); (4) emergency admissions; (5) the patients who transferred from other hospitals; (6) pregnancy or lactation

We collected the following data through the hospital big data query and analysis system:

1. Basic information: gender, age, height, weight, medical insurance, etc.
2. Clinical information: admission paths, admission time, admission departments, discharge time, discharge unit, length of stay, mode of payment；
3. Disease Information: admission diagnosis, disease coding at admission, the first discharge diagnosis, the coding of first discharge diagnosis, the second discharge diagnosis, the third discharge diagnosis, outcome (recovery, improvement, not cured, death, transfer to another hospital)
4. Operation information: surgical name, surgery code,
5. oral nutritional supplement: drug names, unit price
6. laboratory examination: hemoglobin, albumin, prealbumin
7. hospitalization costs: total cost, self-pay cost, other cost, the type of medical insurance； Researchers will compare ONS group to see the clinical outcomes and health economic impact.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18 years old;
2. length of hospital stay ≥3days;
3. Only ONS was used as enteral nutrition or no enteral nutrition was received.

Exclusion Criteria:

1. age<18;
2. length of hospital stay<3 days;
3. the patients who received enteral nutrition other than ONS (such as tube feeding); (4) emergency admissions;

(5) the patients who transferred from other hospitals; (6) pregnancy or lactation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: hospitalized patients with nutritional risk
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2023-10-07 (Estimated); Primary Completion 2023-11-07 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
total cost | through study completion, an average of 1 month
  The total cost of hospitalization for the patient

SECONDARY OUTCOMES:
mortality | through study completion, an average of 1 month
  the number of deaths during the hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided